CLINICAL TRIAL: NCT04656418
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-arm Study to Investigate the Efficacy and Safety of Subcutaneous Administration of CSL312 (Garadacimab) in the Prophylactic Treatment of Hereditary Angioedema
Brief Title: CSL312 (Garadacimab) in the Prevention of Hereditary Angioedema Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSL312_3001; 2020-000570-25 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-07 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSL312 (Experimental): Participants received a CSL312 loading dose of 400 mg as two 200 mg SC injections in Month 1 along with CSL312 of 200 mg subcutaneous (SC) injections, once monthly from Months 2 to 6.
  Interventions: Biological: CSL312
- Placebo (Placebo Comparator): Participants received a CSL312 matched loading dose of placebo as two SC injections in Month 1 along with CSL312 matched placebo SC injections, once monthly from Months 2 to 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSL312 — Fully human immunoglobulin G subclass 4/lambda recombinant monoclonal antibody
  Other Names: Factor XIIa inhibitor monoclonal antibody; garadacimab
  Arms: CSL312
Drug: Placebo — Buffer without active ingredient
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled, parallel-arm study to investigate the efficacy and safety of subcutaneous administration of CSL312 (garadacimab) in the prophylactic treatment of hereditary angioedema.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 12 years of age; diagnosed with clinically confirmed C1-INH hereditary angioedema; experience ≥ 3 attacks during the 3 months before screening.

Note: For subjects taking any prophylactic HAE therapy during the 3 months before Screening, ≥ 3 HAE attacks may be documented over 3 consecutive months before commencing the prophylactic therapy.

Exclusion Criteria:

* Concomitant diagnosis of another form of angioedema such as idiopathic or acquired angioedema, recurrent angioedema associated with urticarial or hereditary angioedema type 3

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring LLC
Locations (28):
- United States (8):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - Raffi Tachdjian MD, Inc., Santa Monica, California
  - Allergy and Asthma Clinical Research, Walnut Creek, California
  - Institute of Asthma and Allergy, Chevy Chase, Maryland
  - Bernstein Clinical Research Center LLC, Cincinnati, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Canada (4):
  - University of Alberta - Research Transition Facility, Edmonton, Alberta
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Gordon Sussman Clinical Research Inc., Toronto, Ontario
  - Clinique specialisee en allergie de la Capitale, Québec
- Germany (5):
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt am Main, Hesse
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Leipzig, Leipzig
  - CRC Clinical Research / Hautklinik und Poliklinik der Universitätsklinik Mainz, Mainz
  - HZRM Hämophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- Semmelweis University, Budapest, Hungary
- Barzilai University Medical Center, Ashkelon, Israel
- Japan (8):
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Kobe University Hospital, Kobe, Hyōgo
  - St.Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa
  - Saitama Medical Center, Saitama, Kawagoe-shi
  - Saga University Hospital, Saga, Saga-shi
  - Koga Community Hospital, Yaizu-shi, Shizuoka
  - Juntendo University Hospital, Bunkyo, Tokyo
  - Saiyu Soka Hospital, Saitama
- Amsterdam UMC, Location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.

REFERENCES:
- [Derived] Craig TJ, Reshef A, Li HH, Jacobs JS, Bernstein JA, Farkas H, Yang WH, Stroes ESG, Ohsawa I, Tachdjian R, Manning ME, Lumry WR, Saguer IM, Aygoren-Pursun E, Ritchie B, Sussman GL, Anderson J, Kawahata K, Suzuki Y, Staubach P, Treudler R, Feuersenger H, Glassman F, Jacobs I, Magerl M. Efficacy and safety of garadacimab, a factor XIIa inhibitor for hereditary angioedema prevention (VANGUARD): a global, multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Apr 1;401(10382):1079-1090. doi: 10.1016/S0140-6736(23)00350-1. Epub 2023 Feb 28. PMID 36868261
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in Canada, Germany, Hungary, Israel, Japan, Netherlands, and the United States from 27 January 2021 to 07 June 2022.
Pre-assignment Details: A total of 80 participants were screened, of which 64 participants were randomized and received the loading dose in the treatment period.
Groups:
- CSL312: Participants received a CSL312 loading dose of 400 mg as two 200 mg subcutaneous (SC) injections in Month 1 along with CSL312 of 200 mg SC injections, once monthly from Months 2 to 6.
Period: Overall Study
Arm/Group | CSL312 | Placebo
Started | 39 | 25
Intention-to-treat (ITT) Analysis Set (ITT analysis set included all the randomized participants who provided written informed consent and underwent study screening procedures.) | 39 | 25
Safety Analysis Set (Safety analysis set included all the randomized participants who provided written informed consent, underwent study screening procedures and received at least 1 dose of the investigational product.) | 39 | 25
Completed | 38 | 22
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all the randomized participants who provided written informed consent and underwent study screening procedures.
Groups:
- CSL312: Participants received a CSL312 loading dose of 400 mg as two 200 mg SC injections in Month 1 along with CSL312 of 200 mg SC injections, once monthly from Months 2 to 6.
- Total: Total of all reporting groups
Arm/Group | CSL312 | Placebo | Total
Number analyzed (Participants) | 39 | 25 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (17.45) | 37.8 (12.80) | 41.2 (15.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 14 | 38
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 37 | 23 | 60
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4 | 2 | 6
  Race: Black or African American | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: White | 33 | 22 | 55
  Race: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 3 | 8
  Netherlands | 2 | 1 | 3
  Hungary | 2 | 0 | 2
  United States | 12 | 9 | 21
  Japan | 4 | 2 | 6
  Israel | 7 | 2 | 9
  Germany | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Time-Normalized Number of Hereditary Angioedema (HAE) Attacks Per Month During Treatment Period
Description: Time-normalized number of HAE attacks per month during treatment was calculated per participant as: [number of HAE attacks / length of participant treatment in days] * 30.4375.
Time Frame: First injection up to 6 months
Population: ITT analysis set included all the randomized participants who provided written informed consent and underwent study screening procedures. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: number of HAE attacks per month
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 24
number of HAE attacks per month | 0.27 (0.683) | 2.01 (1.341)
Statistical Analysis 1: Comparison: CSL312 vs Placebo; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Compared the time-normalized number of HAE attacks in the active and placebo arms by using a two-sided Wilcoxon test (Hierarchical Testing H01) at alpha = 5%

2. Secondary Outcome: Percentage Change in the Time-normalized Number of HAE Attacks Per Month During the Treatment Period Compared to the Run-in Period
Description: Percentage change in the time-normalized number of HAE attacks was calculated within a participant as:
  100 * [1 - (time-normalized number of HAE attacks per month during treatment period / time-normalized number of HAE attacks per month during run-in period)]. Time-normalized number of HAE attacks per month during treatment period was calculated per participant as: [number of HAE attacks / length of participant treatment in days] * 30.4375.
Time Frame: 6 months, first 3-months and second 3-months of treatment period
Population: ITT analysis set included all the randomized participants who provided written informed consent and underwent study screening procedures. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: percentage change in HAE attacks/month
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 24
percentage change in HAE attacks/month
  6 Months of Treatment | 90.67 (22.433) | 20.21 (42.661)
  First 3-months of Treatment | 91.10 (21.255) | 18.89 (53.837)
  Second 3-months of Treatment: number analyzed (Participants) | 39 | 22
  Second 3-months of Treatment | 90.12 (25.624) | 29.87 (55.529)
Statistical Analysis 1: Comparison: CSL312 vs Placebo; 6 Months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Compared the time-normalized number of HAE attacks in the active and placebo arms by using a two-sided Wilcoxon test

3. Secondary Outcome: Time-Normalized Number of HAE Attacks Per Month Requiring On-Demand Treatment
Description: Time-normalized number of HAE attacks per month requiring on-demand treatment was calculated per participant as: [number of HAE attacks requiring on-demand treatment / length of participant in days] * 30.4375.
Time Frame: 6 months, first 3-months and second 3-months of treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of HAE attacks per month
Units Other Than Participants: Total number of HAE attacks
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 24
Number analyzed (Total number of HAE attacks) | 63 | 264
number of HAE attacks per month
  6 Months of Treatment | 0.23 (0.663) | 1.86 (1.412)
  First 3-months of Treatment: number analyzed (Total number of HAE attacks) | 31 | 144
  First 3-months of Treatment | 0.24 (0.748) | 1.76 (1.378)
  Second 3-months of Treatment: number analyzed (Participants) | 39 | 22
  Second 3-months of Treatment: number analyzed (Total number of HAE attacks) | 32 | 120
  Second 3-months of Treatment | 0.23 (0.610) | 1.80 (1.626)
Statistical Analysis 1: Comparison: CSL312 vs Placebo; 6 Months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Tested the differences between the active and placebo arms using a two-sided Wilcoxon test at alpha = 5%
Statistical Analysis 2: Comparison: CSL312 vs Placebo; First 3-months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Tested the differences between the active and placebo arms using a two-sided Wilcoxon test at alpha = 5%
Statistical Analysis 3: Comparison: CSL312 vs Placebo; Second 3-months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Tested the differences between the active and placebo arms using a two-sided Wilcoxon test at alpha = 5%

4. Secondary Outcome: Time-Normalized Number of Moderate or Severe HAE Attacks Per Month
Description: Time-normalized number of moderate or severe HAE attacks per month during treatment period was calculated per participant as: [number of moderate or severe HAE attacks / length of participant treatment in days] * 30.4375.
Time Frame: 6 months, first 3-months and second 3-months of treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of HAE attacks per month
Units Other Than Participants: Total number of HAE attacks
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 24
Number analyzed (Total number of HAE attacks) | 63 | 264
number of HAE attacks per month
  6 Months of Treatment | 0.13 (0.296) | 1.35 (1.166)
  First 3-months of Treatment | 0.12 (0.305) | 1.25 (1.091)
  Second 3-months of Treatment: number analyzed (Participants) | 39 | 22
  Second 3-months of Treatment | 0.13 (0.320) | 1.24 (1.296)
Statistical Analysis 1: Comparison: CSL312 vs Placebo; 6 Months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Tested the differences between the active and placebo arms using a two-sided Wilcoxon test at alpha = 5%
Statistical Analysis 2: Comparison: CSL312 vs Placebo; First 3-months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Tested the differences between the active and placebo arms using a two-sided Wilcoxon test at alpha = 5%
Statistical Analysis 3: Comparison: CSL312 vs Placebo; Second 3-months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Tested the differences between the active and placebo arms using a two-sided Wilcoxon test at alpha = 5%

5. Secondary Outcome: Time-normalized Number of HAE Attacks Per Month in the First 3-months and Second 3-months of Treatment Period
Description: as for outcome 1
Time Frame: First 3-months and second 3-months of treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of HAE attacks per month
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 24
number of HAE attacks per month
  First 3-months of Treatment | 0.26 (0.749) | 1.97 (1.287)
  Second 3-months of Treatment: number analyzed (Participants) | 39 | 22
  Second 3-months of Treatment | 0.28 (0.652) | 1.86 (1.603)
Statistical Analysis 1: Comparison: CSL312 vs Placebo; First 3-months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Tested the differences between the active and placebo arms using a two-sided Wilcoxon test at alpha = 5%
Statistical Analysis 2: Comparison: CSL312 vs Placebo; Second 3-months of treatment; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Tested the differences between the active and placebo arms using a two-sided Wilcoxon test at alpha = 5%

6. Secondary Outcome: Relative Difference in Means in the Time-Normalized Number of HAE Attacks Per Month Between CSL312 to Placebo
Description: Relative difference in means in the time-normalized number of HAE attacks per month CSL312 to Placebo was calculated as: 100 * [(mean time-normalized number of HAE attacks for CSL312 - mean time-normalized number of HAE attacks for placebo) / mean time-normalized number of HAE attacks for placebo]. Time-normalized number of HAE attacks per month during treatment was calculated per participant as: [number of HAE attacks / length of participant treatment in days] * 30.4375.
Time Frame: 6 months, first 3-months and second 3-months of treatment period
Population: ITT analysis set included all randomized participants who provided written informed consent and underwent study screening procedures. 'Overall number of participants analyzed' indicates number of participants with data available for outcome measure (OM) analysis. 'Number analyzed' indicates number of participants with data available for analysis at specified time point. As pre-specified in protocol and SAP, data for this OM was reported for participants of CSL312 and Placebo Comparison group.
Measure: Mean (95% Confidence Interval); unit: number of HAE attacks per month
Groups:
- CSL312 and Placebo Comparison Group: CSL312: Participants received a CSL312 loading dose of 400 mg as two 200 mg SC injections in Month 1 along with CSL312 of 200 mg SC injections, once monthly from Months 2 to 6.
  Placebo: Participants received a CSL312 matched loading dose of placebo as two SC injections in Month 1 along with CSL312 matched placebo SC injections, once monthly from Months 2 to 6.
Arm/Group | CSL312 and Placebo Comparison Group
Number analyzed (Participants) | 63
number of HAE attacks per month
  6 Months of Treatment | -86.51 [-95.68 to -57.84]
  First 3-months of Treatment | -86.64 [-95.87 to -56.76]
  Second 3-months of Treatment: number analyzed (Participants) | 61
  Second 3-months of Treatment | -85.01 [-95.62 to -48.74]
Statistical Analysis 1: Comparison: CSL312 and Placebo Comparison Group; Test type: Other — Test for differences; p < 0.001, Two-sided Wilcoxon test — Compared the time-normalized number of HAE attacks in the active and placebo arms by using a two-sided Wilcoxon test (Hierarchical testing H02) at alpha = 5%

7. Secondary Outcome: Percentage of Participants With a Response to Subject's Global Assessment of Response to Therapy (SGART)
Description: SGART is a self-assessment by the participant and measures the subject's overall treatment response to the investigational product using the following ratings: 0 (none: worse or no response at all, not acceptable), 1 (poor: very little response, not acceptable), 2 (fair: some response, acceptable but could be better), 3 (good: good response, acceptable), and 4 (excellent: excellent response, as good as can be imagined).
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 38 | 24
percentage of participants
  None | 2.6 | 41.7
  Poor | 7.9 | 16.7
  Fair | 7.9 | 8.3
  Good | 15.8 | 20.8
  Excellent | 65.8 | 12.5

8. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE), Serious Adverse Event (SAE), and AEs of Special Interest (AESI)
Description: AE is any untoward medical occurrence in a participant administered with an investigational product which does not necessarily have a causal relationship with treatment, can be any unfavorable and unintended sign, symptom, or disease temporally associated with use of an investigational product, whether or not considered related to product. SAE is any untoward medical occurrence that results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, is a congenital anomaly or birth defect, or is a medically significant event. An AESI is an AE of scientific and medical concern specific to sponsor's product or program, for which ongoing monitoring and rapid communication by investigator to sponsor is appropriate.
Time Frame: From first dose of study drug up to 3 months after the last injection (approximately 8 months)
Population: Safety analysis set included all the randomized participants who provided written informed consent, underwent study screening procedures and received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 25
Participants
  AE | 25 | 15
  SAE | 1 | 0
  AESI | 0 | 0

9. Secondary Outcome: Number of Participants With CSL312-induced Anti-CSL312 Antibodies
Time Frame: Up to 8 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 25
Participants | 1 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Assessments Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Laboratory assessments included: Hematology, biochemistry, urinalysis, and coagulation parameters.
Time Frame: From first dose of study drug up to 3 months after the last injection (approximately 8 months)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 25
Participants | 1 | 2

11. Secondary Outcome: Percentage of Participants With at Least One AE, SAE, and AESI
Description: as for outcome 8
Time Frame: From first dose of study drug up to 3 months after the last injection (approximately 8 months)
Population: Safety analysis set included all the randomized participants who provided written informed consent, underwent study screening procedures and received at least 1 dose of the investigational product. The percentage of participants are rounded off to the single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 25
percentage of participants
  AE | 64.1 | 60.0
  SAE | 2.6 | 0
  AESI | 0 | 0

12. Secondary Outcome: Percentage of Participants With CSL312-induced Anti-CSL312 Antibodies
Time Frame: Up to 6 months
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 25
percentage of participants | 2.6 | 0

13. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormalities in Laboratory Assessments Reported as TEAEs
Description: Laboratory assessments included: Hematology, biochemistry, urinalysis, and coagulation parameters.
Time Frame: From first dose of study drug up to 3 months after the last injection (approximately 8 months)
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | CSL312 | Placebo
Number analyzed (Participants) | 39 | 25
percentage of participants | 2.6 | 8.0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 3 months after the last injection (approximately 8 months)
Description: Safety analysis set included all the randomized participants who provided written informed consent, underwent study screening procedures and received at least 1 dose of the investigational product.
Arm/Group | CSL312 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/39 | 0/25
Other Adverse Events (participants affected / at risk) | 17/39 | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CSL312 (N=39) | Placebo (N=25)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CSL312 (N=39) | Placebo (N=25)
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
COVID-19 (Infections and infestations) | 0 | 3
Gastrointestinal infection (Infections and infestations) | 2 | 1
Conjunctivitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Fatigue (General disorders) | 0 | 3
Injection site erythema (General disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 2
Headache (Nervous system disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Visual impairment (Eye disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT04656418/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT04656418/SAP_001.pdf